CLINICAL TRIAL: NCT06098937
Title: Orientation Characteristics of Kalifilcon A Daily Disposable Toric Contact Lenses Compared to Commercially Available Daily Disposable Toric Contact Lenses
Brief Title: Kalifilcon A Toric Compared to Commercially Available Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ROC-23-007
Record Dates: First submitted 2023-09-29; First posted 2023-10-25 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Astigmatism
Keywords: Contact Lens
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Kalifilcon A Daily Disposable Toric (Experimental): Kalifilcon A Daily Disposable Toric
  Interventions: Device: Kalifilcon Toric Lens
- Total1 for Astigmatism (Active Comparator): Total1 for Astigmatism
  Interventions: Device: Total1 for Astigmatism
- Precision1 for Astigmatism (Active Comparator): Precision1 for Astigmatism
  Interventions: Device: Precision1 for Astigmatism
- MyDay Toric (Active Comparator): MyDay Toric
  Interventions: Device: MyDay Toric

INTERVENTIONS:
Device: Kalifilcon Toric Lens — Kalifilcon A Daily Disposable Toric for Ametropia
  Arms: Kalifilcon A Daily Disposable Toric
Device: Total1 for Astigmatism — Total1 for Astigmatism
  Arms: Total1 for Astigmatism
Device: Precision1 for Astigmatism — Precision1 for Astigmatism
  Arms: Precision1 for Astigmatism
Device: MyDay Toric — MyDay Toric
  Arms: MyDay Toric

SUMMARY:
Approximately thirty contact lens adapted subjects will be enrolled in this feasibility, bilateral, randomized, double masked (subject and investigator masked), repeated measures insertion study.

DETAILED DESCRIPTION:
Approximately 30 soft toric contact lens adapted subjects will be enrolled in this feasibility, bilateral, randomized, double masked (subject and investigator masked), repeated measures insertion study. All subjects will be seen for a Screening/Dispensing Visit at which informed consent will be obtained and eligibility will be assessed. If study eligibility is met, subjects will have lenses inserted in random, successive order. Subjects will be receiving each of the study lens types once, in a randomized order. The subject will wear each of the study contact lenses for approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older on the date the Informed Consent Form (ICF) is signed and have capacity to read, understand and provide written voluntary informed consent.
2. Have physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
3. Have no active ocular disease or allergic conjunctivitis.
4. Not be using any topical ocular medications.
5. Be willing and able to follow instructions.
6. Have signed a statement of informed consent.

Exclusion Criteria:

1. Participating in a conflicting study in the opinion of the Investigator.
2. Considered by the Investigator to not be a suitable candidate for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bausch & Lomb, Incorporated, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Kalifilcon A Daily Disposable Toric Compared to Total1, Precision1, and MyDay Toric.: Participants received kalifilcon A daily disposable toric, commercially available Total1 for Astigmatism, Precision1 for Astigmatism, and MyDay Toric.
Period: Overall Study
Arm/Group | Kalifilcon A Daily Disposable Toric Compared to Total1, Precision1, and MyDay Toric.
Started | 30
Kalifilcon A Daily Disposable Toric | 30
Total1 for Astigmatism | 30
Precision1 for Astigmatism | 30
MyDay Toric Lenses | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Kalifilcon A Daily Disposable Toric, Total1, Precision1, and MyDay Toric.: Participants received kalifilcon A daily disposable toric, Total1 for Astigmatism, Precision1 for Astigmatism, and MyDay Toric.
Arm/Group | Kalifilcon A Daily Disposable Toric, Total1, Precision1, and MyDay Toric.
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age 28 to 70 | 46.6 (12.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Primary Gaze Orientation for 5 Minutes
Description: Primary gaze orientation is measured in degrees using a slit lamp and reticule.
Time Frame: 5 minutes after lens insertion
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Kalifilcon A Daily Disposable Toric: Participants received kalifilcon A daily disposable toric
- Total1 for Astigmatism: Participants received commercially available Total1 for Astigmatism
- Precision1 for Astigmatism: Participants received Precision1 for Astigmatism
- MyDay Toric: Participants received MyDay Toric
Arm/Group | Kalifilcon A Daily Disposable Toric | Total1 for Astigmatism | Precision1 for Astigmatism | MyDay Toric
Number analyzed (Participants) | 30 | 30 | 30 | 30
degrees | 3.3 (5.19) | 2.8 (4.16) | 2.4 (3.96) | 3.6 (5.45)

ADVERSE EVENTS:
Time Frame: throughout study, average of 22 days
Description: There were no Adverse Events
Groups:
- Kalifilcon A Daily Disposable Toric, Total1, Precision1, and MyDay Toric.: Participants received kalifilcon A daily disposable toric, commercially available Total1 for Astigmatism, Precision1 for Astigmatism, and MyDay Toric.
Arm/Group | Kalifilcon A Daily Disposable Toric, Total1, Precision1, and MyDay Toric.
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT06098937/Prot_SAP_000.pdf